CLINICAL TRIAL: NCT05476029
Title: Study on Exosomes and Biomarkers in Plasma and Alveolar Lavage Fluid of Patients With Sepsis Complicated With ARDS
Brief Title: Changes of Exosomes and Biomarkers in Plasma and Alveolar Lavage Fluid of Patients With Sepsis Complicated With ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor, Tianjin Nankai Hospital
Other Study IDs: NKYY_YXKT_IRB_2022_018_01
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Sepsis Complicated With ARDS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Within 24h after admission to ICU, blood samples and alveolar lavage fluid were collected and transferred to a cleaning tube and stored in a refrigerator at -80°C for exosome sorting and identification, differential miRNAs, and analysis of serum oxidation and inflammatory indicators
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis complicated with ARDS group: Blood samples and alveolar lavage fluid were collected within 24h after admission to ICU. After blood samples were collected, they were placed in static stratification at 4°C and centrifuged at 3000×g for 10 min. Serum samples and alveolar lavage fluid samples were transferred to a cleaning tube and stored in a refrigerator at -80°C for exosome sorting, identification, differential miRNAs, and analysis of serum oxidation and inflammatory indicators.
  Interventions: Diagnostic Test: Blood samples and alveolar lavage fluid were collected
- control group: Blood samples and alveolar lavage fluid were collected. After blood samples were collected, they were placed in static stratification at 4°C and centrifuged at 3000×g for 10 min. Serum samples and alveolar lavage fluid samples were transferred to a cleaning tube and stored in a refrigerator at -80°C for exosome sorting, identification, differential miRNAs, and analysis of serum oxidation and inflammatory indicators.
  Interventions: Diagnostic Test: Blood samples and alveolar lavage fluid were collected

INTERVENTIONS:
Diagnostic Test: Blood samples and alveolar lavage fluid were collected — Blood samples and alveolar lavage fluid were collected for exosome sorting and identification, differential miRNAs, and analysis of serum oxidation and inflammatory indicators.

SUMMARY:
In this study, serum samples and alveolar lavage fluid from patients with sepsis complicated with ARDS were studied. The differential miRNAs of inflammatory exosomes in patients with sepsis lung injury were screened, and Sestrin2, HO-1 and PPARγ proteins, oxidative stress and inflammatory indexes in serum and alveolar lavage fluid were measured simultaneously, to explore the relationship between HO-1, oxidative inflammatory indexes and metabolic indexes. These results provide an important reference for assisting the management of ARDS disease and predicting the adverse outcomes of sepsis patients with ARDS.

DETAILED DESCRIPTION:
1. Title: Study on exosomes and biomarkers in plasma and alveolar lavage fluid of patients with sepsis complicated with ARDS
2. Research center: monocentric
3. The Design of the study: Randomized, double-blind
4. The population of the study: 1)Age ≥18, no gender or ethnic limitation. 2) Patients with sepsis who meet the criteria of sepsis -3 and ARDS is defined according to Berlin standard.
5. Interventions: Within 24h after admission to ICU, blood samples and alveolar lavage fluid were collected and transferred to a cleaning tube and stored in a refrigerator at -80°C for exosome sorting and identification, differential miRNAs, and analysis of serum oxidation and inflammatory indicators.

7. The aim of the research: to explore the relationship between HO-1, oxidative inflammatory indexes and metabolic indexes and provide an important reference for assisting the management of ARDS disease and predicting the adverse outcomes of sepsis patients with ARDS.

8. Outcome： Differential miRNAs of inflammatory exosomes were screened from patients with septic lung injury, and ho-1, PPARγ or other positive indicators were used to regulate differential miRNAs 9. The estimated duration of the study：2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old；
2. Patients with sepsis who meet the criteria for sepsis -3；
3. Agree to participate in this study and sign informed consent；

Exclusion Criteria:

1. Refuse to participate in this study；
2. Patients with left atrial hypertension to prevent the inclusion of patients with abnormal oxygenation index due to cardiogenic pulmonary edema；
3. Pregnant or lactation patients
4. Patients are currently being enrolled in another study
5. The attending physician or researcher considers that there are other circumstances (reasons to be noted) that are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis meeting the criteria of sepsis -3 and complicating lung injury
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Differential miRNAs of inflammatory exosomes were screened from patients with septic lung injury | 1year
  Differential miRNAs of inflammatory exosomes were screened from patients with septic lung injury, and ho-1, PPARγ or other positive indicators were used to regulate differential miRNAs.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD,PhD, Study Chair — Tianjin Nankai Hospital
Locations (1):
- Plasma and alveolar lavage fluid, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang D, Wang X, Si M, Yang J, Sun S, Wu H, Cui S, Qu X, Yu X. Exosome-encapsulated miRNAs contribute to CXCL12/CXCR4-induced liver metastasis of colorectal cancer by enhancing M2 polarization of macrophages. Cancer Lett. 2020 Apr 1;474:36-52. doi: 10.1016/j.canlet.2020.01.005. Epub 2020 Jan 10. PMID 31931030
- [Result] Rezaei R, Baghaei K, Amani D, Piccin A, Hashemi SM, Asadzadeh Aghdaei H, Zali MR. Exosome-mediated delivery of functionally active miRNA-375-3p mimic regulate epithelial mesenchymal transition (EMT) of colon cancer cells. Life Sci. 2021 Mar 15;269:119035. doi: 10.1016/j.lfs.2021.119035. Epub 2021 Jan 13. PMID 33450254
- [Result] Kalluri R, LeBleu VS. The biology, function, and biomedical applications of exosomes. Science. 2020 Feb 7;367(6478):eaau6977. doi: 10.1126/science.aau6977. PMID 32029601
- [Result] Chekanova JA, Gregory BD, Reverdatto SV, Chen H, Kumar R, Hooker T, Yazaki J, Li P, Skiba N, Peng Q, Alonso J, Brukhin V, Grossniklaus U, Ecker JR, Belostotsky DA. Genome-wide high-resolution mapping of exosome substrates reveals hidden features in the Arabidopsis transcriptome. Cell. 2007 Dec 28;131(7):1340-53. doi: 10.1016/j.cell.2007.10.056. PMID 18160042
- [Result] Wu X, Liu Z, Hu L, Gu W, Zhu L. Exosomes derived from endothelial progenitor cells ameliorate acute lung injury by transferring miR-126. Exp Cell Res. 2018 Sep 1;370(1):13-23. doi: 10.1016/j.yexcr.2018.06.003. Epub 2018 Jun 5. PMID 29883714
- [Result] Zhou Y, Li P, Goodwin AJ, Cook JA, Halushka PV, Chang E, Zingarelli B, Fan H. Exosomes from endothelial progenitor cells improve outcomes of the lipopolysaccharide-induced acute lung injury. Crit Care. 2019 Feb 13;23(1):44. doi: 10.1186/s13054-019-2339-3. PMID 30760290
- [Result] Shin CH, Byun J, Lee K, Kim B, Noh YK, Tran NL, Park K, Kim SH, Kim TH, Oh SJ. Exosomal miRNA-19a and miRNA-614 Induced by Air Pollutants Promote Proinflammatory M1 Macrophage Polarization via Regulation of RORalpha Expression in Human Respiratory Mucosal Microenvironment. J Immunol. 2020 Dec 1;205(11):3179-3190. doi: 10.4049/jimmunol.2000456. Epub 2020 Oct 28. PMID 33115854
- [Result] Zheng L, Su J, Zhang Z, Jiang L, Wei J, Xu X, Lv S. Salidroside regulates inflammatory pathway of alveolar macrophages by influencing the secretion of miRNA-146a exosomes by lung epithelial cells. Sci Rep. 2020 Nov 27;10(1):20750. doi: 10.1038/s41598-020-77448-6. PMID 33247202